CLINICAL TRIAL: NCT03009383
Title: Efficacy of a Bedside Portable Endoscopy on Identifying the Esophageal Foreign Body
Brief Title: A Bedside Portable Endoscopy for the Esophageal Foreign Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KNUH20161227
Record Dates: First submitted 2016-12-26; First posted 2017-01-04 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Esophageal Foreign Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A bedside portable endoscopy (Experimental)
  Interventions: Device: A bedside portable endoscopy

INTERVENTIONS:
Device: A bedside portable endoscopy

SUMMARY:
The purpose of this study is to determine whether a bedside portable endoscopy is effective in identifying the esophageal foreign body in the emergency room.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visit the emergency room due to apparent foreign body in esophagus

Exclusion Criteria:

* Patients unable to insert a portable endoscopy through the nasal cavity
* Patients unable to undergo conventional esophagogastroduodenoscopy for a gold standard examination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value of the bedside portable endoscopy to identify esophageal foreign body defined by comparison with conventional esophagogastroduodenoscopy as a gold standard method | Within 1 hr after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi JH, Choi JH, Lee YJ, Lee HK, Choi WY, Kim ES, Park KS, Cho KB, Jang BK, Chung WJ, Hwang JS. Comparison of a novel bedside portable endoscopy device with nasogastric aspiration for identifying upper gastrointestinal bleeding. World J Gastroenterol. 2014 Jul 7;20(25):8221-8. doi: 10.3748/wjg.v20.i25.8221. PMID 25009396